CLINICAL TRIAL: NCT05760885
Title: Multisensory Augmentation to Improve the Standing Balance of People With Chronic Stroke
Brief Title: Multisensory Augmentation for Post-stroke Standing Balance
Acronym: MAB
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A4545-R; I01RX004545 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a Control or an Experimental group. The Experimental group will receive sensory augmentation during balance training, while the Control group will not.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not be informed of which group participants are assigned to, and will not be present during an training sessions. As participants will be aware whether or not they will receive sensory augmentation (in the form of vibration), they can not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensory Augmentation (Experimental): Participants will receive sensory augmentation in the form of non-invasive vibration, while balance training is performed as described below.
  Interventions: Behavioral: Balance training with sensory augmentation
- Control (Active Comparator): Participants will receive balance training, without any sensory augmentation.
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Balance training with sensory augmentation — Participants will complete 20 balance training sessions, in which they are required to keep their balance while standing on a platform that translates under their feet. During training, sensory augmentation will be delivered with an intensity controlled in real-time by their center of pressure motion. The difficulty of the balance training task will progressively increase over successive training sessions.
  Arms: Sensory Augmentation
Behavioral: Balance training — Participants will complete 20 balance training sessions, in which they are required to keep their balance while standing on a platform that translates under their feet. During training, no sensory stimulation will be delivered. The difficulty of the balance training task will progressively increase over successive training sessions.
  Arms: Control

SUMMARY:
Many individuals who experience a stroke have problems with their balance. In part, these balance problems may be due to sensory issues. This study will test whether sensory augmentation has the potential to improve post-stroke balance. Sensory augmentation is a method by which non-invasive vibration is used to enhance the sensory information available to users, which may make it easier to feel where they are and prevent losses of balance.

DETAILED DESCRIPTION:
The objective of this study is to design a novel multisensory augmentation approach to improve the control of standing balance in people with chronic stroke. With sensory augmentation, artificial feedback provides the nervous system with information about the dynamic state of the body, which can be used to prevent losses of balance. This clinical trial will investigate whether multisensory augmentation produces sustained balance improvements when applied as a training device. These potential improvements will be assessed by comparing the results of clinical and biomechanical assessments before and after a 10-week balance training program, in which half of the participants will be randomly assigned sensory augmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 21 years;
2. Experience of a stroke at least 6 months prior to participation;
3. Berg Balance Scale score less than 52
4. Ability to stand independently for at least 1 minute without wearing an AFO or other brace that would preclude delivery of stimulation to the ankle or foot sole
5. Provision of informed consent

Exclusion Criteria:

1. Resting blood pressure higher than 220/110 mm Hg
2. History of unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living
3. Pre-existing neurological disorders or dementia
4. Severe visual impairment
5. History of DVT or pulmonary embolism within 6 months
6. Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale score change | Before and after a 10-week period of balance training
  A standard clinical assessment to measure balance performance during various functional tasks

SECONDARY OUTCOMES:
Limits of Stability score (paretic direction) | Before and after a 10-week period of balance training
  A standard assessment of how far participants are willing and able to shift their weight toward the paretic leg while standing
Limits of Stability score (non-paretic direction) | Before and after a 10-week period of balance training
  A standard assessment of how far participants are willing and able to shift their weight toward the non-paretic leg while standing
Mediolateral center of pressure displacement | Before and after a 10-week period of balance training
  A measure of sideways sway, which will be quantified as participants stand on a platform that translates sideways, challenging participant balance
Mediolateral center of pressure velocity | Before and after a 10-week period of balance training
  A measure of sideways sway, which will be quantified as participants stand on a platform that translates sideways, challenging participant balance

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C. Dean, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified data that contains no protected participant information. This data will be shared in the form of pre-prints and through online servers upon study results publication.
Supporting Information: Study Protocol, ICF
Time Frame: We will share de-identified data upon study results publication, which we anticipate will happen within one year after study completion. Data will remain available in perpetuity.
Access Criteria: All consumers of the scientific literature will have access to the shared de-identified data.